CLINICAL TRIAL: NCT03255993
Title: Multiple Doses Study to Evaluate the Tolerability and Pharmacokinetics of SPH3127 in Chinese Healthy People
Brief Title: The Tolerability and Pharmacokinetics of Multiple Doses of SPH3127 in Chinese Healthy People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPH3127-102
Record Dates: First submitted 2017-08-08; First posted 2017-08-21 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — SPH3127

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- SPH3127 100mg (Experimental): A single dose of SPH3127 50 mg*2 qd *7 days
  Interventions: Drug: SPH3127 50mg
- Placebo to SPH3127 100mg (Placebo Comparator): A single dose of placebo matching to SPH3127 50mg*2 qd *7 days
  Interventions: Drug: Placebo matching to SPH3127 50mg
- SPH3127 200mg (Experimental): A single dose of SPH3127 100 mg*2 qd *7 days
  Interventions: Drug: SPH3127 100mg
- Placebo to SPH3127 200mg (Placebo Comparator): A single dose of placebo matching to SPH3127 100mg*2 qd *7 days
  Interventions: Drug: Placebo matching to SPH3127 100mg
- SPH3127 400mg (Experimental): A single dose of SPH3127 100 mg*4 qd *7 days
  Interventions: Drug: SPH3127 100mg
- Placebo to SPH3127 400mg (Placebo Comparator): A single dose of placebo matching to SPH3127 100mg*4 qd *7 days
  Interventions: Drug: Placebo matching to SPH3127 100mg

INTERVENTIONS:
Drug: SPH3127 50mg — SPH3127 50mg
  Other Names: SPH3127 is a new study drug for hypertension
  Arms: SPH3127 100mg
Drug: SPH3127 100mg — SPH3127 100mg
  Other Names: SPH3127 is a new study drug for hypertension
  Arms: SPH3127 200mg; SPH3127 400mg
Drug: Placebo matching to SPH3127 50mg — Placebo matching to SPH3127 50mg
  Other Names: Placebo is oral tablet to matching to SPH3127 50mg
  Arms: Placebo to SPH3127 100mg
Drug: Placebo matching to SPH3127 100mg — Placebo matching to SPH3127 100mg
  Other Names: Placebo is oral tablet to matching to SPH3127 50mg
  Arms: Placebo to SPH3127 200mg; Placebo to SPH3127 400mg

SUMMARY:
This study was a single center, parallel, randomized, double blind, placebo-controlled phase Ib clinical trial to to evaluate the safety and tolerability and pharmacokinetics of SPH3127 tablet in healthy subjects by increasing multiple dosing

DETAILED DESCRIPTION:
Three panels(100mg, 200mg, 400mg), each consisting of eight participants (The number of individual subjects in each group was not less than 1/3 of the total number).Participants begin to receive the first dose of SPH3127 100mg. Then Participants begin to receive the second dose of SPH3127 200mg,after the researchers confirmed that the 100mg dose group was safe and well tolerated.Then the third dose of SPH3127 400mg must wait for the result of the second dose's safety and tolerability. If the subjects during escalating dose to the biggest tolerate dose group were not well tolerated, the study must adjust the maximum dose group and fall to a low dose group to conduct another test.

ELIGIBILITY:
Inclusion Criteria:

1. The body mass index is 18-28kg/m2 (including the critical value), which allows the minimum weight of men to be 50kg (including the critical value) and 45kg for women (including the critical value).
2. Before the study,participant has know about the significance , potential benefits, inconveniences and potential risks of the study
3. Participant has understood the research's procedure and sign the informed consent .

Exclusion Criteria:

* Participant who are Pregnancy, lactating women, and planned trials begin within six months of pregnancy
* Participant who has abnormal Physical examination, laboratory examination results and clinical significance (such as: liver function examination - aspartate aminotransferase (AST) and alanine aminotransferase (ALT) more than 1.5 times that of the upper limit of normal)
* Participant who has a history of cardiovascular, liver, kidney, digestive tract, nervous system, blood system, familial hematologic disease, abnormal thyroid function, or mental abnormality
* Participant who has drug allergy history and anaphylactic reaction
* Participant who took oral contraceptive in 6 months
* Participant who used any drug (including Chinese herbal medicine) within 1 week.
* Participant who donated blood within 2 months
* Participant who participated clinical trials of any drug in 3 months (as subjects)
* Participant who has any positive result of virus serology check: human immunodeficiency virus antigen antibody (HIV Ag/Ab) and hepatitis c virus (HCV) - immunoglobulin G(IgG) antibody to IgG, hepatitis b surface antigen (HBsAg) and treponema pallidum antibody (TP)
* Participant who are used to smoke, alcohol abuse, eat coffee and strong tea and drug abuse
* Participant who the researchers believe that there are volunteers who are not suitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Baseline to 13-16 days post last dose
  to assess incidence and intensity of Adverse Events according to Common Toxicity Criteria (CTC version 4.03) associated with increasing doses of SPH3127

SECONDARY OUTCOMES:
Plasma area under curve (AUC)(0-∞) of SPH3127 | 10 minutes predose, 0.17hour, 0.33hour, 0.5hour, 0.75hour, 1hour, 1.25hour, 1.5hour, 2hour, 4hour, 6hour, 8hour, 12hour postdose at Day 1 and 7; 10 minutes predose at Day 2; 10 minutes predose, 1hour postdose at Day 5 or 6
  to evaluate Plasma AUC(0-∞) of SPH3127
Change from baseline in laboratory hematology values | Baseline to 13-16 days post last dose
  to evaluate the Change from baseline in laboratory hematology values
Change from baseline in laboratory chemistry values | Baseline to 13-16 days post last dose
  to evaluate the Change from baseline in laboratory chemistry values
Change from baseline in laboratory urinalysis values | Baseline to 13-16 days post last dose
  to evaluate the Change from baseline in laboratory urinalysis values
Change from baseline in ECG | Baseline to 13-16 days post last dose
  to evaluate the Change from baseline in ECG
Maximum Plasma Concentration (Cmax) of SPH3127 | 10 minutes predose, 0.17hour, 0.33hour, 0.5hour, 0.75hour, 1hour, 1.25hour, 1.5hour, 2hour, 4hour, 6hour, 8hour, 12hour postdose at Day 1 and 7;10 minutes predose at Day 2; 10 minutes predose, 1hour postdose at Day 5 or 6
  to evaluate Plasma Cmax of SPH3127
Plasma Maximum time to peak (Tmax) of SPH3127 | 10 minutes predose, 0.17hour, 0.33hour, 0.5hour, 0.75hour, 1hour, 1.25hour, 1.5hour, 2hour, 4hour, 6hour, 8hour, 12hour postdose at Day 1 and 7;10 minutes predose at Day 2; 10 minutes predose, 1hour postdose at Day 5 or 6
  to evaluate Plasma Tmax of SPH3127
Apparent terminal half-life of SPH3127 | 10 minutes predose, 0.17hour, 0.33hour, 0.5hour, 0.75hour, 1hour, 1.25hour, 1.5hour, 2hour, 4hour, 6hour, 8hour, 12hour postdose at Day 1 and 7;10 minutes predose at Day 2; 10 minutes predose, 1hour postdose at Day 5 or 6
  to evaluate terminal half-life of SPH3127

CONTACTS AND LOCATIONS:
Locations (1):
- The capital medical university affiliated Beijing anzhen hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Jing S, Xu R, Yang K, Liu W, Zhang L, Ke Y, Xia G, Lin Y. Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SPH3127: A Phase I, Randomized, Double-Blind, Placebo-Controlled Trial. Clin Ther. 2021 Apr;43(4):735.e1-735.e14. doi: 10.1016/j.clinthera.2021.01.025. Epub 2021 Feb 27. PMID 33653620